CLINICAL TRIAL: NCT00278304
Title: A Pilot Study of MR-Guided High Dose Rate Brachytherapy With MR Image Acquisition for Patients With Cervical Cancer
Brief Title: Radiation Therapy in Treating Patients With Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000454997; NCI-05-C-0233; NCT00214396 (obsolete NCT alias)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2006-04

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Radiotherapy

INTERVENTIONS:
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving external-beam radiation together with internal radiation works in treating patients with cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of magnetic resonance-guided, endocavitary, high-dose rate brachytherapy implants in patients with stage IB-IVB cervical cancer.
* Provide more reliable dose-volume estimations based on three-dimensional imaging-based treatment planning in patients treated with this regimen.

Secondary

* Determine the toxic effects and treatment tolerance in patients treated with this regimen.
* Correlate three-dimensional dose-volume histograms of organs at risk with treatment toxicity in patients treated with this regimen.
* Determine the disease status, time and patterns of relapse, and survival of patients treated with this regimen.

OUTLINE: Patients undergo external beam radiotherapy 4-5 days a week for up to 7 weeks. Patients also undergo MRI-guided high-dose brachytherapy comprising one brachytherapy implant a week for 3-6 implants. Brachytherapy may be administered during or after external beam radiotherapy.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the cervix of 1 of the following cellular subtypes:

  * Squamous cell
  * Adenocarcinoma
  * Adenosquamous cell
* Stages IB-IVA disease

  * Stage IVB disease allowed provided the impact on the quality of life is tremendous (e.g., "frozen pelvis" or massive pelvic disease and fistula formation, severe pain, or bleeding)
* Measurable and/or evaluable disease on MRI

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* No physical or physiological capacity that would preclude study treatment
* No cognitively impaired patients who cannot provide informed consent
* Not pregnant or nursing
* Negative pregnancy test
* No contraindication to MRI, including any of the following:

  * Weight > 136 kg
  * Allergy to MR contrast agent
  * Pacemakers, cerebral aneurysm clips, shrapnel injury, or implantable electronic devices
* No significant unrelated systemic illness
* No serious infections
* No significant cardiac, pulmonary, hepatic, or other organ dysfunction that would preclude study treatment
* Must be medically fit to receive anesthesia

PRIOR CONCURRENT THERAPY:

* No prior definitive brachytherapy procedures

  * Ring implants or intravaginal cones for the relief of excessive bleeding allowed
* No prior definitive surgical oncologic procedures (e.g., radical hysterectomy)
* Concurrent chemotherapy, immunotherapy, or hormonal therapy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-09; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Feasibility
Comparison of dose-volume estimations based on 3D imaging-based treatment planning, with the traditional point dose method based on orthogonal radiographs

SECONDARY OUTCOMES:
Tolerance
Toxicity
Correlate three-dimensional dose-volume histograms of organs at risk with treatment toxicity
Disease status
Time and patterns of relapse
Survival distributions

CONTACTS AND LOCATIONS:
Overall Officials: Shervin Karimpour, MD, Principal Investigator — NCI - Radiation Oncology Branch; ROB
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States